CLINICAL TRIAL: NCT03685383
Title: Cytokine Adsorption in Post-cardiac Arrest Syndrome in Patients Requiring Extracorporeal Cardiopulmonary Resuscitation
Acronym: CYTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Daniel Duerschmied, Prof. Dr. (Associate Professor), University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYTER_SC_2018
Record Dates: First submitted 2018-09-05; First posted 2018-09-26 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Cardiac Arrest; Extracorporeal Circulation; Extracorporeal Membrane Oxygenation; Cytokine Storm; Cytokine Release Syndrome; Post-Cardiac Arrest Syndrome
Keywords: Extracorporeal Circulation; Extracorporeal Membrane Oxygenation; Cytokine Adsorption; Post-Cardiac Arrest Syndrome; Cardiac Arrest; Cardio-Pulmonary Resuscitation
MeSH Terms: conditions — Heart Arrest; Cytokine Release Syndrome; Post-Cardiac Arrest Syndrome

STUDY DESIGN:
Intervention Model Description: two-groups (treatment vs. control), pseudo-randomized, monocentric, nonblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group: eCPR + CytoSorb (Experimental): In addition to standard treatment in patients undergoing eCPR in the intervention group the CytoSorb removal column will be added to the ECLS-system (intervention: CytoSorb removal column in eCPR).
  Interventions: Device: Cytosorb removal column in eCPR
- control group: eCPR - CytoSorb (Active Comparator): Patients in the control group will receive standard treatment established for eCPR patients on our ICU. This standard treatment includes, among others, targeted temperature management (TTM) for the first 72 hours. For the use of ECLS as well as TTM we are following well established standard operating procedures (control: standard eCPR (va-ECMO)).
  Interventions: Device: standard eCPR (va-ECMO)

INTERVENTIONS:
Device: Cytosorb removal column in eCPR — In addition to standard treatment in eCPR in the study group a CytoSorb removal column is added to the va-ECMO system for the prevention of post-cardiac arrest syndrome.
  Arms: intervention group: eCPR + CytoSorb
Device: standard eCPR (va-ECMO) — Standard treatment in eCPR with a established va-ECMO system.
  Arms: control group: eCPR - CytoSorb

SUMMARY:
Almost all patients with refractory cardiac arrest, who are primarily stabilized under ongoing cardiopulmonary resuscitation by transcutaneous implantation of a venoarterial extracorporeal membrane oxygenation system (va-ECMO for eCPR) develop post-cardiac arrest syndrome (PCAS). PCAS is characterised by cytokine storm resulting in vasodilation and membrane leakage, which is poorly controlled and often fatal. Case reports and data from the investigators' single-center registry indicate that cytokine adsorption with the CytoSorb removal column can be safely added to va-ECMO, but its efficacy and safety have not been examined systematically. This pilot study will assign all comers undergoing eCPR to va-ECMO with or without cytokine adsorber in a 1:1 fashion. This will ensure comparability and allow analysing clinical endpoints, but is limited by sample size (according to their experience the investigators expect approximately 20 cases per year). The investigators will however be able to generate important data about safety, secondary endpoints such as Interleukin-6-removal or vasopressor use and low-power data about efficacy concerning the primary endpoint 30-day survival.

DETAILED DESCRIPTION:
Survival after out-of-hospital cardiac arrest (OHCA) as well as intra-hospital cardiac arrest (IHCA) is poor and remains on low levels over the past decades. Introduction of eCPR has promised to improve survival, however, so far there is no supporting data for this claim. In a recent registry study at the investigators' hospital they determined survival rates of 8.5% (OHCA) and 18.9% (IHCA), respectively. Almost all patients with refractory cardiac arrest, who are primarily stabilized under ongoing cardiopulmonary resuscitation by transcutaneous implantation of a veno-arterial extracorporeal membrane oxygenation system (va-ECMO for eCPR) develop post-cardiac arrest syndrome (PCAS). PCAS is characterised by cytokine storm resulting in vasodilation and membrane leakage, which is poorly controlled and often fatal. Case reports and data from the investigators' single-center registry indicate that cytokine adsorption with the CytoSorb removal column can be safely added to va-ECMO, but its efficacy and safety have not been examined systematically.

First, the investigators aim to assess the influence of treatment with the CytoSorb removal column over 72 hours after cardiac arrest and resuscitation using eCPR on 30-day-survival. As secondary endpoints, the investigators will assess the efficacy of Interleukin-6-removal, vasopressor-use and fluid-substitution, the latter two as a subsidiary of the degree of PCAS. Finally, the investigators will asses the safety of the use of the CytoSorb column in eCPR/va-ECMO.

The investigators hypothesize that the use of the CytoSorb column in eCPR/va-ECMO is a safe and efficient means to manage the consequences of PCAS and thus reduce 30-day mortality after eCPR.

All patients admitted to the investigators' hospital after successful CPR and implantation of va-ECMO/ ECLS (extracorporeal life support, eCPR) will be included in the trial. In a 1:1 manner participants will be assigned to the intervention and control groups.

Experimental intervention:

In addition to standard treatment in patients undergoing eCPR in the intervention group the CytoSorb removal column will be added to the ECLS-system.

Control intervention:

Patients in the control group will receive standard treatment established for eCPR patients on our ICU. This standard treatment includes, among others, targeted temperature management (TTM) for the first 72 hours. For the use of ECLS as well as TTM we are following well established standard operating procedures.

Duration of intervention per patient:

The duration of the intervention will be 72 hours. Each CytoSorb removal column can be used for 24 hours, so all patients in the intervention group will receive 3 subsequent filters during the study period.

Follow-up per patient:

The follow-up period for each patient in the trial will be 30 days.

Key inclusion criteria:

All patients admitted to our ICU after successful CPR undergoing eCPR will be included in the trial.

Key exclusion criteria:

The single exclusion criteria for the trial is, if decision has been made before admission to our ICU to terminate treatment within the next 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to our ICU after successful CPR undergoing eCPR will be included in the trial.

Exclusion Criteria:

* The single exclusion criteria for the trial is, if decision has been made before admission to our ICU to terminate treatment within the next 24 hours.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
survival after 30 days | 30 days
  rate of survival after 30 days after eCPR

SECONDARY OUTCOMES:
secondary outcome measure: cytokine-clearance | 72 hours
  Interleukin-6 level (patient blood)
secondary outcome measure: vasopressor use | 72 hours
  vasopressor-use (µg/h/kg bodyweight)
secondary outcome measure: fluid substitution | 72 hours
  fluid substitution (ml/h/kg bodyweight)
secondary outcome measure: renal function | 72 hours
  serum creatinin level
secondary outcome measure: serum-lactate | 72 hours
  serum-lactate level

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Duerschmied, Prof. Dr., Principal Investigator — University of Freiburg
Locations (1):
- University Clinic Freiburg, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Supady A, Zahn T, Kuhl M, Maier S, Benk C, Kaier K, Bottiger BW, Bode C, Lother A, Staudacher DL, Wengenmayer T, Duerschmied D. Cytokine adsorption in patients with post-cardiac arrest syndrome after extracorporeal cardiopulmonary resuscitation (CYTER) - A single-centre, open-label, randomised, controlled trial. Resuscitation. 2022 Apr;173:169-178. doi: 10.1016/j.resuscitation.2022.02.001. Epub 2022 Feb 7. PMID 35143902